CLINICAL TRIAL: NCT07181941
Title: Pharmacodynamically Monitored Linvoseltamab Dosing De-Escalation in Relapsed Multiple Myeloma
Brief Title: Response-Based Dose Reduction of Linvoseltamab in the Treatment of Relapsed, Refractory, or Triple-Class Relapsed/Refractory Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RG1125714; NCI-2025-06211 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-09-12; First posted 2025-09-19 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Multiple Myeloma; Refractory Multiple Myeloma; Triple-Class Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Biopsy; Magnetic Resonance Spectroscopy; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Step-up dosing (linvoseltamab) (Experimental): Patients receive linvoseltamab IV over 30-240 minutes QW in weeks 1-14 and then Q2W thereafter in the absence of disease progression or unacceptable toxicity. Patients are evaluated for disease response starting at week 3 and continuing every 4 weeks. Patients without VGPR or better continue receiving linvoseltamab IV over 30-240 minutes Q2W in the absence of disease progression or unacceptable toxicity. Patients who do achieve VGPR or better after a minimum of 14 weeks of therapy are then assigned to 1 of 3 dose de-escalation cohorts. Patients undergo bone marrow aspiration and biopsy and collection of blood samples throughout the trial. Patients may undergo CT or PET/CT throughout the trial if indicated.
  Interventions: Biological: Linvoseltamab; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Biospecimen Collection
- Cohort 1 (Q4W linvoseltamab) (Experimental): Patients receive linvoseltamab IV over 30-240 minutes Q4W in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow aspiration and biopsy and collection of blood samples throughout the trial. Patients may undergo CT or PET/CT throughout the trial if indicated.
  Interventions: Biological: Linvoseltamab; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Biospecimen Collection
- Cohort 2 (Q8W linvoseltamab) (Experimental): Patients receive linvoseltamab IV over 30-240 minutes Q8W in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow aspiration and biopsy and collection of blood samples throughout the trial. Patients may undergo CT or PET/CT throughout the trial if indicated.
  Interventions: Biological: Linvoseltamab; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Biospecimen Collection
- Cohort 3 (Q12W linvoseltamab) (Experimental): Patients receive linvoseltamab IV over 30-240 minutes Q12W in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow aspiration and biopsy and collection of blood samples throughout the trial. Patients may undergo CT or PET/CT throughout the trial if indicated.
  Interventions: Biological: Linvoseltamab; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Biospecimen Collection

INTERVENTIONS:
Biological: Linvoseltamab — Given IV
  Other Names: Anti-BCMA x Anti-CD3 Bispecific Antibody REGN5458; Anti-BCMA/CD3 Bispecific Antibody REGN5458; BCMA x CD3 Bispecific Antibody REGN5458; Linvoseltamab-gcpt; Lynozyfic; REGN 5458; REGN-5458; REGN5458
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This phase I/II trial evaluates the safety and feasibility of early, response-based dose reduction of linvoseltamab in the treatment of patients multiple myeloma that has come back after a period of improvement (relapsed), that does not respond to treatment (refractory), or that is resistant to three classes of therapeutic agents, including proteasome inhibitors, immunomodulatory agents, and monoclonal antibodies (triple-class relapsed/refractory). Linvoseltamab is a bispecific antibody. Upon administration, linvoseltamab binds to the BCMA protein on cancer cells and the CD3 protein on T cells (a type of immune cell). This generates an immune response that stimulates the T cells to kill the cancer cells. Optimal dosing schedules of linvoseltamab have not yet been determined. Reducing the dosage of linvoseltamab may reduce treatment-related side effects while maintaining long-term disease outcomes.

DETAILED DESCRIPTION:
OUTLINE:

STEP-UP DOSING: Patients receive linvoseltamab intravenously (IV) over 30-240 minutes once a week (QW) in weeks 1-14 and then once every 2 weeks (Q2W) thereafter in the absence of disease progression or unacceptable toxicity. Patients are evaluated for disease response starting at week 3 and continuing every 4 weeks. Patients without very good partial response (VGPR) or better continue receiving linvoseltamab IV over 30-240 minutes Q2W in the absence of disease progression or unacceptable toxicity. Patients who do achieve VGPR or better after a minimum of 14 weeks of therapy are then assigned to 1 of 3 dose de-escalation cohorts. Patients undergo bone marrow aspiration and biopsy and collection of blood samples throughout the trial. Patients may undergo computed tomography (CT) or positron emission tomography (PET)/CT throughout the trial if indicated.

COHORT 1: Patients receive linvoseltamab IV over 30-240 minutes once every 4 weeks (Q4W) in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow aspiration and biopsy and collection of blood samples throughout the trial. Patients may undergo CT or PET/CT throughout the trial if indicated.

COHORT 2: Patients receive linvoseltamab IV over 30-240 minutes once every 8 weeks (Q8W) in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow aspiration and biopsy and collection of blood samples throughout the trial. Patients may undergo CT or PET/CT throughout the trial if indicated.

COHORT 3: Patients receive linvoseltamab IV over 30-240 minutes once every 12 weeks (Q12W) in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow aspiration and biopsy and collection of blood samples throughout the trial. Patients may undergo CT or PET/CT throughout the trial if indicated.

After completion of study treatment, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years. Myeloma is not seen in the younger age group and safety of B-cell maturation antigen (BCMA) T-cell engagers (TCE) in this group is not known
* Ability to understand and willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of potential study participants
* Confirmed diagnosis of active multiple myeloma (MM) by International Myeloma Working Group (IMWG) diagnostic criteria
* Patients must have myeloma that is measurable and response evaluable according to 2016 IMWG response criteria. Measurable disease is defined as one of the following, documented ≤ 14 days prior to registration:

  * Serum M protein ≥ 1 g/dl
  * Urine M protein ≥ 200 mg/24h
  * Free light chain (FLC) assay with involved FLC ≥ 10 mg/dl and abnormal FLC ratio
  * A patient with immunoglobulin A (IgA) MM without measurable M protein may be enrolled if quantitative (quant) IgA level ≥ 400 mg/dl and can be followed longitudinally
  * Plasmacytoma target lesion defined as measurable based on at least 1 soft tissue lesion ≥ 2 cm in long axis on CT or PET/CT, if not previously irradiated
  * Skin lesions ≥ 2 cm in long axis as measured with a ruler
* Patients with relapsed or refractory myeloma who have received at least 4 prior lines of therapy including proteasome inhibitor (PI), immunomodulatory imide drug (IMiD), and anti-CD38 monoclonal antibody
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Adequate organ function (based on testing ≤14 days prior to registration):

  * Adequate hematologic function before dosing as measured by:

    * Platelet count ≥50 x 10⁹/L. A patient may not have received a platelet transfusion ≤7 days in order to meet this platelet eligibility requirement
    * Absolute neutrophil count (ANC) ≥1.0 x 10⁹/L. A patient may not have received granulocyte colony stimulating factor (G-CSF) ≤2 days in order to meet this absolute neutrophil count eligibility requirement
    * Hemoglobin ≥8.0 g/dL
  * Adequate renal and hepatic function, defined as:

    * Total bilirubin ≤1.5 x ULN
    * Transaminase (alanine aminotransferase [ALT], aspartate aminotransferase [AST]) ≤2.5 x ULN
    * Alkaline phosphatase ≤2.5 x ULN

      * Patients with Gilbert syndrome do not need to meet this total bilirubin requirement provided that the total bilirubin is unchanged from the baseline value
    * Serum creatinine clearance by Cockcroft-Gault ≥30 mL/min. A patient with a creatinine clearance by Cockcroft-Gault who does not meet eligibility criteria may be considered for enrollment per principal investigator discretion if a measured creatinine clearance (based on 24-hour urine collection or other reliable method) is ≥30 mL/min
* Prior treatment with BCMA-targeted antibody-drug conjugates (ADCs) is allowable if all adverse events (AEs) attributable to these therapies have resolved to grade 1 or lower
* Willing and able to comply with clinic visits and study-related procedures and provide informed consent signed by study patient

Exclusion Criteria:

* Diagnosis of known plasma cell leukemia, known primary systemic light-chain amyloidosis (excluding myeloma-associated amyloidosis), known Waldenström macroglobulinemia (lymphoplasmacytic lymphoma), or known POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Patients with known MM brain lesions or meningeal involvement
* History of known neurodegenerative condition, central nervous system (CNS) movement disorder, or patients with a history of seizure within 12 months prior to study enrollment
* Continuous systemic corticosteroid treatment with more than 10 mg per day of prednisone or anti-inflammatory equivalent within 72 hours of start of study drug
* Live or live attenuated vaccines with replicating potential within 28 days prior to first study drug administration
* Previous treatment with chimeric antigen receptor (CAR) T therapy or any gene therapy products
* Any infection requiring hospitalization or treatment with intravenous (IV) anti-infectives within 2 weeks of first administration of study drug
* Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B (HBV), or hepatitis C (HCV)
* Known allergy or hypersensitivity to components of linvoseltamab (REGN5458)
* Women of childbearing potential (WOCBP) with a positive serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test are ineligible for this study

  * WOCBP are defined as women who are fertile following menarche until becoming postmenopausal, unless permanently sterile. Post-menopausal state is defined as no menses for 12 months without an alternate medical cause
* Participants who are receiving other investigational agents
* Women of childbearing potential (WCOBP) and men who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 6 months after the last dose
* Uncontrolled or concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Another malignancy in the past 5 years, except for non-melanoma skin cancer that has undergone potentially curative therapy or in situ cancer, or any other tumor that has been deemed to be effectively treated with definitive local control and with curative intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects who experience early disease progression | Within 3 months of initiation of dosing de-escalation

SECONDARY OUTCOMES:
Measurable residual disease (MRD) negativity | One year after treatment initiation
  MRD negativity will be assessed at 10e^-6.

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Dhodapkar, MBBS, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No